CLINICAL TRIAL: NCT06267417
Title: Evaluation of The Effect of Low Level Laser Therapy in The Prevention of Chemotherapy Induced Oral Mucositis in Children With Hematological Cancers
Brief Title: Laser Therapy Effect as Preventive Measure for Oral Mucositis in Children With Hematological Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Cancer Hospital Egypt 57357 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CCHE-AML-4/2023
Record Dates: First submitted 2023-07-24; First posted 2024-02-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-02

CONDITIONS: Oral Mucositis
Keywords: low level laser therapy; oral mucositis
MeSH Terms: conditions — Stomatitis | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The outcome evaluator will be a single personnel from the oncology team following up with the case
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser (Experimental): 21 patients will receive Low Level Laser therapy using the wavelength (660 nm) to provide biostimulation at 44 different points in the oral cavity along with the standard preventive protocol in the hospital.
  Interventions: Device: Laser therapy
- Placebo (Sham Comparator): 21 patients will receive a mock treatment which is the exact repetition of the treatment modality but without any laser emission beside the standard preventive protocol applied in the hospital.
  Interventions: Device: Mock treatment

INTERVENTIONS:
Device: Laser therapy — - Laser will be applied with the specified wave length using Diode laser (Sirrolaser Blue ™, USA) device over 5 consecutive days from start of chemotherapy cycle beside the standard preventive protocol applied in the hospital
  Arms: Laser
Device: Mock treatment — The exact repetition of the treatment modality but without any laser emission beside the standard preventive protocol applied in the hospital
  Arms: Placebo

SUMMARY:
Introduction:

Among the most drastic complications of chemotherapy is oral mucositis(OM). It is a painful inflammatory, often ulcerative condition and may increase risk for systemic infections leading to prolonged hospital stays and interruptions of treatment protocol. Many treatment modalities have been introduced for the prevention and treatment of oral mucositis , of which low level laser therapy(LLLT) is gaining popularity. The use of LLLT as a prophylactic treatment for chemotherapy induced oral mucositis in pediatric cancer patients is still lacking robust evidence. Also, the parameters used have not been optimized and no standard method has yet been established. Based on this point, this study will compare photobiomodulation to the conventional preventive program of oral mucositis applied in 57357 children's cancer hospital foundation to determine which will be optimal for the prophylaxis of chemotherapy-induced OM.

Aim:

To assess the effectiveness of low level laser therapy in the prophylaxis of oral mucositis in pediatric patients diagnosed with Hematological cancers.

Methods:

This study is a randomized, prospective, double-blinded trial that will include acute Myeloid leukemia patients admitted to receive chemotherapy cycle between the age of 3 and 18years. These patients will be randomized into two groups: group 1 will receive low level laser therapy and group 2 will receive mock treatment. Patient will be followed to asses the development of oral mucositis on prespecified time points.

DETAILED DESCRIPTION:
This study is a randomized, prospective, double-blinded trial ( patient & outcome assessor) that will include acute Myeloid leukemia patients admitted to receive chemotherapy cycle between the age of 3 and 18years. These patients will be randomized by the Clinical Epidemiology unit using a computer-based method into two groups.

Group I: will receive Low Level Laser Therapy by Diode laser (Sirrolaser Blue ™, USA) at 44 different points in the oral cavity for 5 consequent days from Day 1 to Day 5 of chemotherapy cycle along with the standard preventive protocol in the hospital.

Group II: will receive a mock treatment which is the exact repetition of the treatment modality but without any laser emission beside the standard preventive protocol applied in the hospital.

All patients will be assessed for oral mucositis grade using NCI-CTCAE scale V4 and WHO score on days 1,5,12,19 and 30 .

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients diagnosed with Acute Myeloid Leukemia.
* Children with a minimum age of 3 years and a maximum 18 years.
* Children with sufficient cooperation to accept the treatment and evaluation periods

Exclusion Criteria:

* Patients with limited mouth openings less than 1 cm, due to difficulty of laser radiation.
* Patients with dysplastic oral lesions.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
To measure incidence of oral mucositis in Laser arm versus Placebo arm. | Oral mucositis will be evaluated on Days 1, 5, 12, 19 and 30.
  Evaluate effectiveness of low level laser therapy for the Prevention of chemo-therapy induced oral mucositis.
To measure grade of oral mucositis in patients receiving laser arm placebo arm. | Oral mucositis will be evaluated on Days 1, 5, 12, 19 and 30.
  Oral mucositis will be graded in accordance with the classification criteria of the World Health Organization (WHO, and the National Cancer Institute scale (NCI - Common Terminology Criteria for Adverse Events, version 4.0) will also be used to compare the results.

CONTACTS AND LOCATIONS:
Overall Officials: Reem Elkady, MSc, Principal Investigator — Misr International University
Locations (1):
- Children Cancer Hospital 57357, Cairo, Egypt